CLINICAL TRIAL: NCT01785056
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety and Efficacy of Intravenous Immunoglobulin Treatment in Patients With Systemic Sclerosis
Brief Title: IVIG Treatment in Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00000052
Record Dates: First submitted 2013-01-28; First posted 2013-02-06 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-01

CONDITIONS: Systemic Sclerosis; Diffuse Scleroderma
Keywords: Systemic Sclerosis; Diffuse Scleroderma; SSc
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Privigen (Experimental): Privigen is a ready-to-use, sterile, 10% protein liquid preparation of polyvalent human immunoglobulin G (IgG) for intravenous administration. Subjects will be given 2 g/kg/month of IVIGfor 6 months. Each dose will be split into 2 to 4 infusions on consecutive days to achieve the total monthly dose.
  Interventions: Biological: Privigen
- Placebo (Albuminar-5) (Placebo Comparator): Albuminar-5 is a sterile solution of albumin obtained from large pools of adult human venous plasma and used as the placebo in this study. Albuminar-5 will be administered by the intravenous route and each dose will be split into 2 to 4 infusions on consecutive days to achieve the total monthly dose.
  Interventions: Biological: Privigen

INTERVENTIONS:
Biological: Privigen — Subjects will receive 2 g/kg/mo of Privigen® for 6 months if randomized to the treatment group.

SUMMARY:
The purpose of this research is to study the effects of Privigen (intravenous immunoglobulin) on the skin in patients with scleroderma. Approximately 24 subjects will take part in this investigator-initiated study at Georgetown University Hospital and Johns Hopkins Hospital. This study will last for one year (12 months). This research is being done because systemic sclerosis can cause severe, progressive organ involvement. The investigators hope this study treatment will improve the outcomes in this disease, including skin, muscle, joint, gastrointestinal, and lung involvement.

DETAILED DESCRIPTION:
The investigators propose a double-blind controlled trial of 24 patients with Privigen® (Immune Globulin Intravenous (Human), 10% liquid treatment) with 3:1 randomization. Subjects with scleroderma will be given 2 g/kg/mo of Privigen® or placebo (Albuminar®-5) for 6 months. Scleroderma is generally a progressive disease, and while the skin does improve with time in some patients, others have progressive disease in spite of aggressive treatment. Also, spontaneous improvement in other organ systems is even less likely. Patients entered into the trial will have failed to respond to standard of care treatment over the past 4 months. Thus, the investigators feel that any actual improvement observed can be attributed to the IVIG treatment. Since this is a pilot study, future larger controlled trials will be necessary to clearly demonstrate the effectiveness, but the investigators are hoping that this study will give us signals that will guide the future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse systemic sclerosis with active skin involvement as defined as a mRSS >12, with no improvement or worsening in the previous 4 months in spite of treatment with methotrexate, cellcept, imuran, or anti-TNF agent;
* 18 years of age or older;
* Disease duration of less than 5 years from the first non-Raynaud's symptom of scleroderma.

Exclusion Criteria:

* Use of more than 10 mg of prednisone, or any dose of cytoxan, d-penicillamine, or rituximab in the last 3 months;
* History of deep vein thrombosis (DVT), stroke, or other thromboembolic phenomenon;
* History of anaphylaxis or other serious reaction to human blood or blood products.
* Absolute IgA deficiency
* A prior receipt of IVIg treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
To study the effects of IVIG on the skin in patients with scleroderma | At the 4 month visit
  The modified Rodnan Skin Score (mRSS) will be used to determine the changes in skin

SECONDARY OUTCOMES:
To determine any toxicity of IVIG in scleroderma | At the 4 month visit
  Laboratory assessments (Complete Blood Count (CBC) including liver and electrolytes with differentiation, Complete Metabolic Profile (CMP) including creatinine, and Coombs test) will be performed monthly to monitor toxicity.
To evaluate the effects of IVIG on pulmonary function | At the 4 month visit
  Pulmonary Function Tests (PFTs) will be performed to determine these changes.
Muscle, joint, and inflammatory parameters | At the 4 month visit
  Done by performing a physical exam

OTHER OUTCOMES:
To study the effects of IVIG on the skin in patients with scleroderma | At the 6 month visit
  The modified Rodnan Skin Score (mRSS) will be used to determine the changes in skin
To determine any toxicity of IVIG in scleroderma | At the 6 month visit
  Laboratory assessments (Complete Blood Count (CBC) including liver and electrolytes with differentiation, Complete Metabolic Profile (CMP) including creatinine, and Coombs test) will be performed monthly to monitor toxicity.
To evaluate the effects of IVIG on pulmonary function | At the 6 month visit
  Pulmonary Function Tests (PFTs) will be performed to determine these changes.
To study the biologic effects of IVIG on gene arrays in skin biopsies | At the 6 month visit
  A skin biopsy will be taken at the Baseline and Month 6 visit to determine the biological effects of IVIG on the skin.
Muscle, joint, and inflammatory parameters | At the 6 month visit
  A physical exam will be performed to determine these changes

CONTACTS AND LOCATIONS:
Overall Officials: Virginia D Steen, MD, Principal Investigator — Georgetown University Hospital
Locations (2):
- United States (2):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland